CLINICAL TRIAL: NCT06083909
Title: Sarcopenic Obesity as Risk Factor for Insulin Resistance in the Elderly
Brief Title: Sarcopenic Obesity in the Elderly
Status: Completed | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00003268
Record Dates: First submitted 2023-10-09; First posted 2023-10-16 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Sarcopenic Obesity; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ageing is associated with progressive and generalized loss of muscle mass and muscle function, also known as Sarcopenia. Increasingly, obesity has become a compounding factor in ageing-related sarcopenia. The coexistence of obesity and sarcopenia is termed sarcopenic obesity (SO). Older adults with SO are at higher risks of developing diabetes, hypertension, stroke, cardiovascular diseases, and cognitive dysfunction than those older adults who suffer from sarcopenia alone or obesity alone. However, there is insufficient information with regard to the interplay between obesity and sarcopenia. The primary objective of this study is to investigate the impact of SO on insulin resistance in people aged 65-85. Our hypothesis is that SO positively influences insulin resistance in the elderly. We propose to investigate sarcopenia and obesity as risk factors for insulin resistance in the geriatric (65-85 years old) population.

ELIGIBILITY:
Inclusion Criteria:

This study will include both male and females aged 65-85 years.

Exclusion Criteria:

1. Lack capacity to consent for the study, or have moderate or severe cognitive impairment;
2. Have difficulty ambulating as evidenced by any one of the following:

   1. Difficulty climbing 10 steps without resting;
   2. Restricted to a wheelchair
3. Have difficulty performing basic activities of daily living;
4. Have had treatment for cancer in the prior 3 years;
5. Have history of cachexia;
6. Have a history of heart failure;
7. Have a permanent pacemaker in situ (due to magnetic resonance scanning);
8. Have an implanted cardioverter-defibrillator (ICD) in situ;
9. Have had myocardial infarction within the last 6 months;
10. Have any of the following chronic health conditions: peripheral arterial disease prostate cancer, rheumatoid arthritis, autoimmune myositis, chronic obstructive pulmonary disease, and asthma;
11. Are receiving therapy with corticosteroids or immunosuppressants.
12. Are taking direct insulin sensitizers (PPAR-gamma agonists, or thiazolidinediones).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The study will include both men and women who are aged 65-85. We plan to recruit a minimum of 25 men and 25 women but no more than 60 of each gender. The maximum sample size is 100. We estimate that less than 10% of the consented participants will not meet the inclusionary criteria and will be withdrawn. As this study involves a solitary study visit, we estimate that less than 5% of the participants will withdraw/be withdrawn/ or be lost to follow up prior to study completion.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
To explore the correlation of sarcopenia and obesity on insulin resistance | 2 years

SECONDARY OUTCOMES:
To explore the correlation between muscle strength and memory loss | 2 years
To explore the correlation of sarcopenic obesity and glucometabolic and cardiovascular risk. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Muthu Periasamy, PhD, Principal Investigator — University of Central Florida; Mariana Dangiolo, MD, Principal Investigator — University of Central Florida; Ali Rizvi, MD, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States